CLINICAL TRIAL: NCT05576116
Title: Combined Bariatric Surgery and Pancreas After Kidney Transplantation for Type II Diabetics
Acronym: ComB-PAK
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-5927
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Pancreas Transplantation

STUDY DESIGN:
Intervention Model Description: The first phase of the study will assign participants (n=10) to undergo Sleeve Gastrectomy (SG) prior to PAK. 3 months post-SG, patients will be activated on the pancreas transplant waitlist.
  If outcomes are favourable, the study may move to phase II (single group, n=10), which would investigate a combined surgery (simultaneous SG and pancreas transplantation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Staggered Approach (Experimental): The first 10 participants enrolled will undergo Sleeve Gastrectomy a minimum of 3 months prior to Pancreas Transplant.
  Interventions: Procedure: Sleeve Gastrectomy AND Pancreas after Kidney Transplantation (Staggered Approach)
- Group 2: Combined Approach (Experimental): Eligible participants will undergo SG and pancreas transplantation simultaneously
  Interventions: Procedure: Combined Sleeve Gastrectomy and Pancreas transplantation

INTERVENTIONS:
Procedure: Sleeve Gastrectomy AND Pancreas after Kidney Transplantation (Staggered Approach) — Participants will undergo sleeve gastrectomy a minimum of 3 months prior to Pancreas Transplant. SG will be performed using the standard technique.
  Pancreas transplant will be performed as per standard procedure.
  Arms: Group 1: Staggered Approach
Procedure: Combined Sleeve Gastrectomy and Pancreas transplantation — Simultaneous SG and pancreas transplantation
  Arms: Group 2: Combined Approach

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of sleeve gastrectomy combined with pancreas after kidney (PAK) transplantation as a means of achieving normoglycemia, insulin independence, reduced insulin resistance, and kidney graft function preservation in the T2DM population. in the first year post pancreas after kidney transplant. Safety and efficacy data will be collected from the time of enrollment until participants reach 1 year post PAK transplant. Data will be compared to historical data from TGH's renal and pancreas transplant programs.

DETAILED DESCRIPTION:
Diabetes is the leading cause of renal dysfunction and failure in Canada. Many patients will require dialysis and some with qualify for and receive a renal transplant. While a renal transplant can restore kidney function in diabetics, it does not address the underlying cause of the kidney disease. Patients remain at high risk of future morbidity from diabetes, including cardiovascular disease, retinopathy, neuropathy, and damage to the new graft. Notably, hyperglycemia is the largest risk factor to the renal bed. Good control of blood glucose levels is essential to minimize these effects but is not easily achieved or maintained.

Pancreas transplantation eliminates the use of exogenous insulin and normalizes glucose levels in the blood. Patients with Type I diabetes are routinely offered Pancreas transplant -either Pancreas After Kidney (PAK) or Simultaneous -pancreas-kidney (SPK). In rare circumstances, patients can also receive a pancreas alone (PTA). At UHN, the investigators have offered SPK transplants to select patients with type II DM who are within weight criteria (BMI <30), but the investigators do not routinely offer PAK transplants to patients with DMII as these patients are overweight and suffering from insulin resistance. Patients with DMII may not be able to achieve normoglycemia and may continue to require exogenous insulin supplementation, after PAK alone.

Weight loss in severely overweight individuals with DMII is known to improve insulin sensitivity. The majority of patients with DM II are overweight and have associated metabolic syndrome. Obesity and metabolic syndrome are themselves major risk factors for poor long-term outcomes in kidney transplantation. Weight loss can lead to improvements in all metabolic syndrome diagnostic criteria, however, it can be difficult to achieve significant and sustained weight loss in the context of insulin resistance associated with DM II. Patients who have already received a kidney transplant have the added metabolic side effects of immunosuppressive medications.

To ensure excellent long-term outcomes with kidney transplantation, it is critically important to investigate strategies to minimize obesity, control diabetes, and improve metabolic and cardiovascular risk factors. Weight loss can be achieved through dieting and exercise, but most patients who diet regain their former weight or gain additional weight. Sleeve gastrectomy (SG) is an aggressive but well-tolerated treatment for obesity which can lessen the risk factors associated with metabolic syndrome and associated poor transplant outcomes.

The investigators hypothesize that combining SG and PAK in patients with DM II who have previously undergone renal transplant will result in improvement of glycemic control, metabolic syndrome criteria, preserved/improved renal graft function and be well tolerated.

This study will investigate the safety and efficacy of SG prior to PAK (staggered approach) compared to simultaneous SG and PAK (combined approach). Safety and efficacy data will be compared to historical data from TGH's renal and pancreas transplant programs. Controls will consist of DMII patients having undergone kidney transplant only, and DMII patients having undergone SPK.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Females must be post-menopausal, surgically sterile or practicing adequate birth control for the duration of the study period
* Recipient of a kidney graft (either live or deceased donor) due to diabetic nephropathy
* Minimum 6 months post-Kidney transplantation surgery
* BMI >30
* Possess 3 of 4 metabolic syndrome components

  * Elevated waist circumference (>88cm for women; >102cm for men)
  * Elevated Triglycerides (>150mg/dL) or drug treatment for elevated triglycerides
  * Low HDL cholesterol (<40mg/dL for men; <50mg/dL for women)
  * Elevated blood pressure (systolic >130mmHg or diastolic >85mmHg) or hypertensive drug treatment
* T2DM - fasting c-peptide of >900 pmol/L
* insulin dependent >1 year

Exclusion Criteria:

* eGFR < 60
* Abnormal alb/cr ratio >2.9
* Cigarette, cigar or pipe smoking; Occasional cannabis smoking is allowable, but not recommended
* Significant peripheral vascular disease that would prevent pancreas from safely being implanted (this is assessed as part of SOC pancreas transplant workup)
* Previous bariatric surgery
* Presence of any other condition that could compromise the patient's ability to safely undergo, or benefit from SG procedure.
* Known BK nephropathy or significant vascular damage to the kidney graft

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients achieving normoglycemia | month 12
  The primary study endpoint will be the proportion of patients who achieve normoglycemia (as defined by HbA1c <6%) by Month 12 post-PAK. This will be compared to the proportion of patients among the historical controls who achieve normoglycemia through medical treatment alone and have undergone kidney transplant alone or simultaneous pancreas-kidney transplantation.

SECONDARY OUTCOMES:
Change in body weight (kg) from baseline to post-SG (group 1); baseline to post-Pancreas Tx M3 (group 2) | month 3
  Change in body weight (kg) from baseline to post-SG (group 1); baseline to post-Pancreas Tx M3 (group 2)
Change in body weight (kg) from baseline to post-PAK | month 12
  Change in body weight (kg) from baseline to post-PAK
Change in HbA1c levels | month 12
  Change in HbA1c levels
Body mass index (BMI) | month 12
  Body mass index (BMI)
Waist circumference | month 12
  Waist circumference
Change in renal graft function post-PAK | months 3,6, 9 and 12
  Change in renal graft function measured by creatinine/urea and Alb/Creatinine ratio
HbA1c levels post-SG | month 3
  HbA1c levels post-SG (group 1)
HbA1c levels post-PAK | months 3,6, 9 and 12
  HbA1c levels post-PAK
Proportion of participants with morbid obesity post PAK | month 12
  Proportion of participants with morbid obesity (defined as BMI > 35) post PAK

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Reichman, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] AlEnazi NA, Ahmad KS, Elsamahy IA, Essa MS. Feasibility and impact of laparoscopic sleeve gastrectomy after renal transplantation on comorbidities, graft function and quality of life. BMC Surg. 2021 May 4;21(1):235. doi: 10.1186/s12893-021-01138-x. PMID 33947375
- [Background] Viscido G, Gorodner V, Signorini FJ, Campazzo M, Navarro L, Obeide LR, Moser F. Sleeve Gastrectomy after Renal Transplantation. Obes Surg. 2018 Jun;28(6):1587-1594. doi: 10.1007/s11695-017-3056-0. PMID 29294221